CLINICAL TRIAL: NCT04160702
Title: Using Virtual Reality to Assess the Efficacy of a Motivational Interviewing Intervention to Increase Bystander Behaviors
Brief Title: Using VR to Assess the Efficacy of a Motivational Interviewing Intervention to Increase Bystander Behaviors
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 19260
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Sexual Assault
Keywords: sexual assault prevention; motivational interviewing; bystander intervention

STUDY DESIGN:
Intervention Model Description: Individuals will be randomly assigned to complete either a motivational interviewing intervention to increase bystander behaviors or an assessment only control condition. The outcome variables are post-treatment bystander behaviors, measured through both self-report measures and a virtual realty assessment of bystander behaviors. The primary analyses will consist of a series of multiple regressions with intervention group (0 = control, 1 = MI training) interacting with each of the moderators to predict post-treatment bystander behaviors (self-reported and B-SAVE).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivate-The-Bystander (Experimental): Participants assigned to the MTB condition arm.
  Interventions: Behavioral: Motivate-The-Bystander (MTB)
- Assessment only control condition (No Intervention): Participants assigned to the assessment only condition arm.

INTERVENTIONS:
Behavioral: Motivate-The-Bystander (MTB) — MTB is a motivational interviewing intervention designed to increase bystander intervention behaviors. During MTB, participants will discuss their knowledge and experiences with bystander intervention. Participants will then create a plan to increase their bystander intervention behaviors in the future. The interviewer will utilize a variety of motivational interviewing techniques to help guide the conversation towards change (e.g., asking questions in an open-ended manner, reflecting participants' personal values).
  Arms: Motivate-The-Bystander

SUMMARY:
With the present project, we will a evaluate a new, motivational interviewing (MI) intervention for increasing bystander behaviors to prevent sexual violence. In the intervention, motivational interviewing will be used to build each participant's unique motivation for engaging in bystander intervention behaviors. To assess the efficacy of the intervention, we will utilize the Bystanders in Sexual Assault Virtual Environments (B-SAVE), a virtual reality measure of bystander behaviors, along with self-report measures examining relevant bystander behaviors and attitudes. We will also examine key moderators of intervention efficacy to provide valuable knowledge (e.g., whom the intervention is most effective for) for further tailoring of the intervention.

DETAILED DESCRIPTION:
This study will provide a comprehensive examination of Motivate-The-Bystander and provide information about whom the intervention is most effective for. Specifically, at T1, participants will be randomly assigned to the MTB condition, a motivational interviewing intervention designed to increase participants' bystander intervention behaviors, or an assessment only control condition. All participants will complete a battery of self-report measures, including our three proposed moderators (gender, alcohol use, and rape myth acceptance). Participants assigned to the MTB condition will also engage in a motivational interviewing intervention designed to build each participant's unique motivation for engaging in bystander intervention behaviors. Approximately two months later, at T2, participants will complete a battery of self-report measures assessing their bystander behaviors and attitudes over the past two months. Then, all participants will complete the B-SAVE, where they provide open ended verbal responses to a series of sexually risky and non-risky interactive scenes they witness in the virtual environment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-25, English speaking

Exclusion Criteria:

* Non English speaking.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Bystander in Sexual Assault Virtual Environment (BSAVE) | Two months after the intervention
  The primary outcome measure consists of participants' open ended verbal responses to a series of sexually risky and non-risky interactive scenes they witness while in the virtual house party.

SECONDARY OUTCOMES:
Bystander Attitudes Scale | Two months after the intervention
  A self-report measure assessing participants' bystander related attitudes.
Bystander Behavior Scale | Two months after the intervention
  A self-report measure assessing participants' actual bystander behaviors over the past two months.
Bystander Efficacy Scale | Two months after the intervention
  A self-report measure assessing participants' confidence in their ability to engage in future bystander behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nebraska Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No